CLINICAL TRIAL: NCT06413108
Title: A Phase 1/2a Single Centre, Randomised, Placebo-controlled, Double-blind, Dose-escalation, Age De-escalation, Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Plasmodium Falciparum Transmission-reducing Activity of Monoclonal Antibody TB31F in Malaria-exposed Malian Adults and Children
Brief Title: Safety, Pharmacokinetics, and Plasmodium Falciparum Transmission-reducing Activity of Monoclonal Antibody TB31F in Mali
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Malaria Research and Training Center, Bamako, Mali (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: TB31F Mali
Record Dates: First submitted 2024-05-03; First posted 2024-05-14 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-09

CONDITIONS: Malaria,Falciparum
Keywords: transmission-reducing; monoclonal antibody
MeSH Terms: conditions — Malaria, Falciparum | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: We will perform two sequential stages of clinical research, each recruiting a distinct cohort of participants to confirm: 1. TB31F safety and 2. TB31F efficacy. The safety cohort will be composed of the three dose groups in adults (groups 1, 2 and 3) and two dose groups in children (groups 4 and 5). The efficacy cohort will be composed of two dose groups in adults and children (group 6). Participants will be randomised within each treatment group to receive a single sub-cutaneous dose of TB31F or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind randomised controlled trial. The treating physician and staff involved with assessing all laboratory outcomes of the study are blinded. The study pharmacist will be unblinded and responsible for randomisation and treatment preparation. Entomology staff involved in the mosquito feeding assays will be blinded for the parasitology results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- 1A: control (Placebo Comparator): 0.2 mL normal saline
  Interventions: Other: Normal saline
- 1B: 10 mg TB31F (Experimental): 0.2 mL (10 mg) TB31F
  Interventions: Drug: TB31F
- 2A: control (Placebo Comparator): 2 mL normal saline
  Interventions: Other: Normal saline
- 2B:100 mg TB31F (Experimental): 2 mL (100 mg) TB31F
  Interventions: Drug: TB31F
- 3A: control (Placebo Comparator): 4 mL normal saline
  Interventions: Other: Normal saline
- 3B: 200 mg TB31F (Experimental): 4 mL (200 mg) TB31F
  Interventions: Drug: TB31F
- 4A: control (Placebo Comparator): 0.2 mL normal saline
  Interventions: Other: Normal saline
- 4B: 10 mg TB31F (Experimental): 0.2 mL (10 mg) TB31F
  Interventions: Drug: TB31F
- 5A: control (Placebo Comparator): 2.0 mL normal saline
  Interventions: Other: Normal saline
- 5B: 100 mg TB31F (Experimental): 2.0 mL (100 mg) TB31F
  Interventions: Drug: TB31F
- 6A: control (Placebo Comparator): 0.6 or 2.0 mL normal saline
  Interventions: Other: Normal saline
- 6B: 30 mg TB31F (Experimental): 0.6 mL (30 mg) TB31F
  Interventions: Drug: TB31F
- 6C: 100 mg TB31F (Experimental): 2.0 mL (100 mg) TB31F
  Interventions: Drug: TB31F

INTERVENTIONS:
Drug: TB31F — transmission-blocking monoclonal antibody TB31F
  Arms: 1B: 10 mg TB31F; 2B:100 mg TB31F; 3B: 200 mg TB31F; 4B: 10 mg TB31F; 5B: 100 mg TB31F; 6B: 30 mg TB31F; 6C: 100 mg TB31F
Other: Normal saline — normal saline as control (placebo)
  Arms: 1A: control; 2A: control; 3A: control; 4A: control; 5A: control; 6A: control

SUMMARY:
Mali faces a significant challenge with malaria, particularly among its younger population. While existing measures like seasonal chemoprevention and vaccination have shown efficacy, further innovations are necessary to combat this disease. The monoclonal antibody TB31F shows promise in reducing the transmission of malaria. This clinical trial will evaluate the safety and efficacy of the monoclonal antibody TB31F.

ELIGIBILITY:
SAFETY COHORT (STUDY ARM 1-5)

Inclusion Criteria:

1. Written/signed informed consent
2. Adult cohorts: 18-50 years of age
3. School-age children cohorts: 10-15 years of age
4. Haemoglobin ≥10 g/dL
5. Non-lactating females of childbearing potential agree to the use of continuous adequate contraception for 28 days after having received investigational product
6. Subject agrees to refrain from blood donation during the study and for 5 months after having received investigational product
7. Subjects are available to attend all study visits
8. In opinion of the investigator, the subject can and will comply with the requirements of the protocol

Exclusion Criteria:

1. Women who are pregnant (tested at baseline and at day 28 after administration of investigational product by urine and/or serum pregnancy testing (β-hCG)) or lactating
2. Symptomatic malaria
3. Current acute or chronic disease, including clinically significant pulmonary, cardiovascular, hepatic, or renal functional abnormality, as determined by history or physical examination
4. Clinically significant abnormal blood chemistries and haematology
5. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 year
6. History of adverse reactions to monoclonal antibodies
7. Administration of immunoglobulin and/or blood products within the three months preceding the first dose of the investigational product or planned administration during the study period
8. Any other condition or situation that would, in the opinion of the investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol

EFFICACY COHORT (STUDY ARM 6)

Inclusion Criteria:

1. Written/signed informed consent
2. 10-50 years of age
3. Haemoglobin ≥10 g/dL
4. Non-lactating females of childbearing potential agree to the use of continuous adequate contraception for 28 days after having received investigational product
5. Subject agrees to refrain from blood donation during the study and for 5 months after having received investigational product
6. Subjects are available to attend all study visits
7. In opinion of the investigator, the subject can and will comply with the requirements of the protocol
8. Asymptomatic P. falciparum mono-infection with asexual parasite densities <3000 parasites/µL
9. Presence of P. falciparum gametocytes on thick blood film at a density >16 gametocytes/µL

Exclusion Criteria:

1. Women who are pregnant (tested at baseline and at day 28 after administration of investigational product by urine and/or serum pregnancy testing (β-hCG)) or lactating
2. Symptomatic malaria
3. Current acute or chronic disease, including clinically significant pulmonary, cardiovascular, hepatic, or renal functional abnormality, as determined by history or physical examination
4. Clinically significant abnormal blood chemistries and haematology
5. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years
6. History of adverse reactions to monoclonal antibodies
7. Administration of immunoglobulin and/or blood products within the three months preceding the first dose of the investigational product or planned administration during the study period
8. Any other condition or situation that would, in the opinion of the investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol
9. Use of anti-malarial drug treatment in the last 14 days
10. Prior receipt of an antimalarial monoclonal antibody
11. Prior receipt of a P. falciparum transmission-blocking vaccine

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 167 (Actual)
Dates: Start 2024-07-12 (Actual); Primary Completion 2026-01-16 (Actual); Study Completion 2026-01-16 (Actual)

PRIMARY OUTCOMES:
Occurrence of at least possibly related solicited local and systemic adverse events | within 7 days of monoclonal antibody TB31F administration
Occurrence of at least possibly related unsolicited adverse events | within 28 days of monoclonal antibody TB31F administration
Occurrence of at least possibly related serious adverse events | from enrollment to the end of follow-up at 28 or 84 days
Terminal serum half-life (t½) of monoclonal antibody TB31F in serum | day 0 [baseline], day 1, day 5, day 7, day 14, day 21, day 28, day 42, day 56, day 84.
Maximum observed serum concentration (Cmax) of monoclonal antibody TB31F in serum | day 0 [baseline], day 1, day 5, day 7, day 14, day 21, day 28, day 42, day 56, day 84.
Time to reach maximum serum concentration (tmax) of monoclonal antibody TB31F in serum | day 0 [baseline], day 1, day 5, day 7, day 14, day 21, day 28, day 42, day 56, day 84.
Accumulation index (Racc) of monoclonal antibody TB31F in serum | day 0 [baseline], day 1, day 5, day 7, day 14, day 21, day 28, day 42, day 56, day 84.
Area under the serum concentration-time curve (AUC0-τ, AUC0-t and AUC) of monoclonal antibody TB31F in serum | day 0 [baseline], day 1, day 5, day 7, day 14, day 21, day 28, day 42, day 56, day 84.
Within-group percent reduction in the proportion of mosquitoes infected at day 5 post-treatment compared to baseline (day 0), assessed through direct membrane feeding assays and measured as oocyst prevalence | day 0 [baseline] & 5

SECONDARY OUTCOMES:
Within-group percent reduction in the proportion of mosquitoes infected in direct skin feeding assay (DSF), compared within groups between baseline and all feeding time points, and between groups at all feeding timepoints. | day 0 [baseline], 1, and 5
Within-group percent reduction in the proportion of mosquitoes infected in direct membrane feeding assays (DMFA), compared within groups between baseline and all feeding time points, and between groups at all feeding timepoints. | day 0 [baseline], 1, 5, and 14
Mosquito infection prevalence, assessed by direct skin feed and measured as the proportion dissected mosquitoes with any number of oocysts, compared within groups between baseline and all feeding time points, and between groups at all feeding timepoints. | day 0 [baseline], 1, and 5
Mosquito infection prevalence, assessed by DMFA and measured as the proportion dissected with any number of oocysts, compared within groups between baseline and all feeding time points, and between groups at all feeding timepoints. | day 0 [baseline], 1, 5, and 14
Mosquito infection intensity, assessed by direct skin feed and measured as the number of oocysts in dissected mosquitoes, compared within groups between baseline and all feeding time points, and between groups at all feeding timepoints. | day 0 [baseline], 1, and 5
Mosquito infection intensity, assessed by DMFA and measured as the average number of oocysts in dissected mosquitoes, compared within groups between baseline and all feeding time points, and between groups at all feeding timepoints. | day 0 [baseline], 1, 5, and 14
Participant infection prevalence, assessed by DSF as the proportion of individuals infectious to any number of mosquitoes, compared within groups between baseline and all feeding time points, and between groups at all feeding timepoints. | day 0 [baseline], 1, and 5
Participant infection prevalence, assessed by DMFA as the proportion of individuals infectious to any number of mosquitoes, compared within groups between baseline and all feeding time points, and between groups at all feeding timepoints. | day 0 [baseline], 1, 5, and 14
Transmission-reducing activity in school-age children and adults, measured as the percent reduction in mean oocyst intensity compared to experimental controls, compared within groups and between groups at all feeding timepoints. | day 0 [baseline], 5, 14, 28, 56, and 84

OTHER OUTCOMES:
Total serum immunoglobulin G level | day 0 [baseline]
  Quantification of the effect of nutritional and protein metabolism status
Serum leptin level | day 0 [baseline]
  Quantification of the effect of nutritional and protein metabolism status
Total protein level | day 0 [baseline]
  Quantification of the effect of nutritional and protein metabolism status
Albumin level | day 0 [baseline]
  Quantification of the effect of nutritional and protein metabolism status
Pre-albumin level | day 0 [baseline]
  Quantification of the effect of nutritional and protein metabolism status
Human genotype analysis at baseline (G6PD, CYP2D6, HBB) | day 0 [baseline]
  To assess human genomic variation in the study population
Plasma biomarkers (i.e. antibodies) at baseline and at post-administration timepoints | day 0 [baseline]
  To assess the presence of plasma biomarkers in the study population
Transmission-blocking activity measured as the percent reduction in mosquito infection prevalence compared to experimental controls, compared within and between groups at all feeding timepoints. | day 0 [baseline], 5, 14, 28, 56, and 84
  To assess the transmission-blocking activity of participant serum after TB31F administration as assessed in the Standard Membrane Feeding Assay (SMFA) at each dose level in adults and school-age children
The concentration of TB31F in serum that provides >80% reduction in the average proportion of infected mosquitoes as measured in direct skin feeding assay after TB31F administration. | day 0 [baseline], 1, and 5.
The concentration of TB31F in serum that provides >80% reduction in the average proportion of infected mosquitoes as measured in direct membrane feeding assays after TB31F administration. | day 0 [baseline], 1, 5, and 14.
The concentration of TB31F in serum that provides >80% transmission blocking activity relative to experimental controls as measured in standard membrane feeding assay after TB31F administration. | day 0 [baseline], 5, 14, 28, 56, and 84
Measure the concentration of TB31F in serum that provides >80% reduction in the average mosquito infection intensity (oocyst number) as measured in direct skin feeding assay after TB31F administration. | day 0 [baseline], 1, and 5.
The concentration of TB31F in serum that provides >80% reduction in the average mosquito infection intensity (oocyst number) as measured in direct membrane feeding assays after TB31F administration. | day 0 [baseline], 1, 5, and 14.
The concentration of TB31F in serum that provides >80% transmission reducing activity relative to experimental controls as measured in standard membrane feeding assay after TB31F administration. | day 0 [baseline], 5, 14, 28, 56, and 84
The correlation between naturally acquired anti-gametocyte immune responses and naturally acquired functional TRA on mosquito infection prevalence, assessed by SMFA and measured as the proportion dissected mosquitoes with any number of oocysts. | day 0 [baseline], 5, 14, 28, 56, and 84
  To assess the impact of naturally acquired TRA, present prior to TB31F administration, on transmission endpoints and TB31F efficacy estimates
The correlation between naturally acquired anti-gametocyte immune responses and naturally acquired functional transmission-reducing activity on mosquito infection intensity, assessed by SMFA and measured as the number of oocysts in dissected mosquitoes. | day 0 [baseline], 5, 14, 28, 56, and 84
  To assess the impact of naturally acquired TRA, present prior to TB31F administration, on transmission endpoints and TB31F efficacy estimates
The correlation between naturally acquired anti-gametocyte immune responses and naturally acquired functional TRA on participant infectivity, assessed by SMFA as the proportion of individuals infectious to any number of mosquitoes. | day 0 [baseline], 5, 14, 28, 56, and 84
  To assess the impact of naturally acquired TRA, present prior to TB31F administration, on transmission endpoints and TB31F efficacy estimates
Parasite genotype analysis (amplicon and whole genome sequencing) | day 0 [baseline]
  To assess human and parasite genomic variation and association with parasite measures
Antibodies and parasite protein in plasma at baseline and at post-administration timepoints | day 0 [baseline], 5, 14, 28, 56, and 84
  To assess the impact of plasma biomarkers on malaria transmission efficiency

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy and Faculty of Medicine and Dentistry, University of Sciences Techniques and Technologies of Bamako, Bamako, Point G, Mali

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, ICF

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-09-30): https://cdn.clinicaltrials.gov/large-docs/08/NCT06413108/SAP_000.pdf